CLINICAL TRIAL: NCT00254748
Title: The Effect of Quetiapine on Psychotic-Like Symptoms in Borderline Personality Disordered Patients: A Randomised Placebo-Controlled Trial
Brief Title: Verkes Borderline Study: The Effect of Quetiapine on Borderline Personality Disordered Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1441C00003
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline personality disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): Flexible doses of 200 mg/day to 600 mg/day quetiapine fumarate
  Interventions: Drug: Quetiapine fumarate

INTERVENTIONS:
Drug: Quetiapine fumarate — flexible doses from 200 mg to 600 mg
  Other Names: Seroquel; 204,636
  Arms: 2
Drug: Placebo — placebo
  Arms: 1

SUMMARY:
In patients with schizophrenia, 'atypical' antipsychotics such as clozapine may be effective in the treatment of psychosis. In patients with borderline personality disorder (BPD), as far as the investigators know, no well designed controlled studies have been performed on the effect of one of the newer atypical antipsychotics on psychotic symptoms.

It is of interest to investigate the benefit of quetiapine treatment in these types of patients. Quetiapine possibly gives less side-effects because of the expected lack of elevated prolactin levels, which is of importance in this patient group, overrepresented by young females. In this double blind, randomized, placebo controlled, 8 week, parallel group, multi-center study, quetiapine (in flexible doses between 200 mg/day and 600 mg/day) will be compared with the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BPD according to Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition (DSM-IV)/Structured Clinical Interview for DSM-IV Axis II Personality Disorders (SCID-II) including criterion 9: transient, stress related paranoid ideation or severe dissociative symptoms.
* In- or outpatients

Exclusion Criteria:

* Depressive disorder
* Bipolar disorder
* Schizoaffective disorder/schizophrenia/delusional disorder/schizotypal personality disorder
* Alcohol- or substance dependence
* Quetiapine doses >100mg od use in the past

Somatic:

* History of trauma capitis
* Visual and auditive disorders
* Neurological disorders (epilepsy)
* Pregnancy
* No adequate contraception
* History of cardial complaints/cardiological disorder
* Known sensitivity for quetiapine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To explore in patients with BPD the effect of quetiapine on psychotic-like symptoms and severity of psychiatric symptoms | assessed at each visit for 8 weeks

SECONDARY OUTCOMES:
To explore the effect of quetiapine on mood, anger, impulsiveness, hostility and anxiety in patients with BPD | assessed at each visit for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (3):
- Netherlands (3):
  - Research Site, Apeldoorn
  - Research Site, Nijmegen
  - Research Site, Veghel

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174